CLINICAL TRIAL: NCT03333746
Title: Phase II Study of Lenalidomide in Combination With Nivolumab In Patients With Relapsed/Refractory Multiple Myeloma
Brief Title: Lenalidomide and Nivolumab in Treating Patients With Relapsed or Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was discontinued due to FDA recommendations of the potential toxicities of the combination of drugs.
Sponsor: Yvonne Efebera (Other)
Collaborators: National Cancer Institute (NCI) (NIH); American Cancer Society, Inc. (Other); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Yvonne Efebera, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-17160; NCI-2017-01653 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA016058 (NIH)
Record Dates: First submitted 2017-10-06; First posted 2017-11-07 (Actual); Results first posted 2019-05-30 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Recurrent Plasma Cell Myeloma; Refractory Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (lenalidomide, nivolumab) (Experimental): Patients receive lenalidomide PO on days 1-21 and nivolumab IV over 1 hour on days 1 and 14. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Lenalidomide; Biological: Nivolumab; Other: Pharmacological Study

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; Revlimid
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase II trial studies how well lenalidomide and nivolumab work in treating patients with multiple myeloma that has come back or does not respond to treatment. Drugs used in chemotherapy, such as lenalidomide, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Monoclonal antibodies, such as nivolumab, may interfere with the ability of cancer cells to grow and spread. Giving lenalidomide and nivolumab may work better in treating patients with multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the efficacy of nivolumab in combination with lenalidomide (Revlimid) in terms of overall response rate in patients with relapse/refractory multiple myeloma (MM).

OUTLINE:

Patients receive lenalidomide orally (PO) on days 1-21 and nivolumab intravenously (IV) over 1 hour on days 1 and 14. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients with evidence of relapse or refractory disease as defined by International Myeloma Working Group (IMWG) criteria and measurable disease as defined by any of the following:

  * Serum m-protein >= 0.5 g/dl (>= 10 g/l)
  * Urine monoclonal protein >= 200 mg/24 hour(h)
  * Involved free light chain (FLC) level >= 10mg/dl (>= 100mg/l) and an abnormal serum free light chain ratio (< 0.26, or > 1.65)
  * Measurable biopsy proven plasmacytoma (should be measured within 28 days of initial investigational agent dosing)
* Patients must have had at least 2 prior line of therapy
* Patients must not have had progression of disease on lenalidomide 25 mg; stable disease on lenalidomide is permitted
* Patient may be enrolled at any time from last line of therapy
* Patients must have absolute neutrophil count (ANC) > 1000/uL
* Platelets >= 75,000/uL, if plasma cell percentage on bone marrow biopsy aspirate or core is > 30%, platelet eligibility requirement will be adjusted to 60,000/ul
* Total bilirubin =< 1.5 mg/dL
* Alkaline phosphatase =< 3 X the upper limit of normal (ULN)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 2 X the ULN
* Patients must have adequate renal function as evidenced by serum creatinine =< 2 mg/dL or calculated creatinine clearance of >= 40 ml/min within 14 days of registration using Modification of Diet in Renal Disease (MDRD) formula
* Patient must be able to swallow capsule or tablet
* Patients must provide informed consent
* Patients must have a left ventricular ejection fraction > 30%, no uncontrolled arrhythmias or New York Heart Association class III-IV heart failure
* Patients must have a Karnofsky performance status >= 70
* A negative pregnancy test will be required for all women of child bearing potential; breast feeding is not permitted
* Fertility requirements

  * Female patients with child bearing potential must have a negative pregnancy test at least 7 days before starting treatment drugs
  * Male patients must agree to use an adequate method of contraception for the duration of the study and for 7 months afterwards
  * Female patients must be either posy-menopausal, free from menses >= 2 years (yrs), surgically sterilized, willing to use two adequate barrier methods of contraception to prevent pregnancy, or agree to abstain from sexual activity starting from screening and for 5 months afterwards
  * Female patients of child bearing potential must agree to comply with the fertility and pregnancy test requirements dictated by the Rev-Assist program

Exclusion Criteria:

* Patients with peripheral neuropathy > Common Terminology Criteria for Adverse Events (CTCAE) grade 2
* Patients receiving concurrent corticosteroids at the time protocol therapy is initiated other than for physiologic maintenance treatment
* History of allergic reaction (including erythema nodosum) to lenalidomide
* Concurrent use of complementary or alternative medicines that would confound the interpretation of toxicities and antitumor activity of the study drugs
* Patients with contraindication to thromboprophylaxis
* Unacceptable cardiac risk factors defined by any of the following criteria: patients with congenital long QT syndrome, any history of ventricular fibrillation or torsade de pointes, bradycardia defined as heart rate (HR) < 50 bpm, left ventricular ejection fraction < 30%
* Patients who have received targeted or investigational agents within 2 weeks or within 5 half-lives of the agent and active metabolites (whichever is longer) and who have not recovered from side effects of those therapies
* Patients who have undergone major surgery =< 2 weeks prior to starting study drug or who have not recovered from the side-effects of surgery
* Patients with known positivity for human immunodeficiency virus (HIV), or hepatitis C; baseline testing for HIV and hepatitis C is not required
* Patients with a history of another primary malignancy that is currently clinically significant or currently requires active intervention, other than non-melanoma skin cancer and carcinoma in situ of the cervix should not be enrolled; patients are not considered to have a ?currently active? malignancy if they have completed therapy for a prior malignancy, are disease free from a prior malignancy for >= 5 yrs and are considered by their physician to be less than 30% risk of relapse
* Patients with active (untreated or relapsed) central nervous system (CNS) metastasis of the patient?s myeloma
* Patients with a history of gastrointestinal surgery or other procedure that might, in the opinion of the investigator(s), interfere with the absorption or swallowing of the study drugs
* Patients with any significant history of non-compliance to medical regimens or unwilling or unable to comply with the instructions given to them by the study staff
* Any other medical condition, including mental illness or substance abuse, deemed by the investigator(s) to likely interfere with the patient?s ability to sign informed consent, cooperate and participate in the study, or interfere with the interpretation of the results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-03-21 (Actual); Primary Completion 2018-08-13 (Actual); Study Completion 2018-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Efebera, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Lenalidomide, Nivolumab)
Started | 1
Completed | 0
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Lenalidomide, Nivolumab)
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: ORR (Overall Response Rate)
Description: Will be assessed by IMWG response criteria. 95% binomial confidence intervals will also be calculated for the estimate of the proportion of responses.
Time Frame: Up to 12 months
Population: data was not collected and analyzed
Arm/Group | Treatment (Lenalidomide, Nivolumab)
Number analyzed (Participants) | 0

2. Secondary Outcome: Overall Survival (OS)
Description: Will evaluate other clinical outcomes using the methods of Kaplan-Meier.
Time Frame: Up to 3 years
Population: data was not collected and analyzed
Arm/Group | Treatment (Lenalidomide, Nivolumab)
Number analyzed (Participants) | 0

3. Secondary Outcome: Progression Free Survival (PFS)
Description: Will evaluate other clinical outcomes using the methods of Kaplan-Meier.
Time Frame: Time from study entry until disease progression or death at trial closure for the per protocol population, assessed up to 3 years
Population: data was not collected and analyzed
Arm/Group | Treatment (Lenalidomide, Nivolumab)
Number analyzed (Participants) | 0

4. Secondary Outcome: Time to Progression (TTP)
Description: Will be assessed.
Time Frame: Time from start of treatment until the date he or she has progression or dies, assessed up to 3 years
Population: data was not collected and analyzed
Arm/Group | Treatment (Lenalidomide, Nivolumab)
Number analyzed (Participants) | 0

5. Other Pre Specified Outcome: Immunomonitoring of Lymphocytes Subsets Including Natural Killer (NK) Cell
Description: Will be explored using graphical analyses as well as summarized quantitatively.
Time Frame: Up to 3 years
Population: data not collected and analyzed
Arm/Group | Treatment (Lenalidomide, Nivolumab)
Number analyzed (Participants) | 0

6. Other Pre Specified Outcome: Immunomonitoring of Lymphocytes Subsets Including T Cell
Description: Will be explored using graphical analyses as well as summarized quantitatively.
Time Frame: Up to 3 years
Population: data not collected and analyzed
Arm/Group | Treatment (Lenalidomide, Nivolumab)
Number analyzed (Participants) | 0

7. Other Pre Specified Outcome: Pharmacokinetics: The Maximum Plasma Concentration (Cmax)
Description: Will be assessed using Cmax for Nivolumab in combination with lenalidomide
Time Frame: Screening, days 1 and 14 of each cycle
Population: data not collected and analyzed
Arm/Group | Treatment (Lenalidomide, Nivolumab)
Number analyzed (Participants) | 0

8. Other Pre Specified Outcome: Pharmacodynamics Profiles:Time to Maximum Plasma Concentration (Tmax)
Description: Will be assessed using Tmax for Nivolumab in combination with lenalidomide
Time Frame: Screening, days 1 and 14 of each cycle
Population: data not collected and analyzed
Arm/Group | Treatment (Lenalidomide, Nivolumab)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse Events were collected up to 8 months during the study was conducted.
Description: Toxicities were assessed according to the NCI Common Terminology Criteria for Adverse Events (CTCAE), Version 4.0.
Arm/Group | Treatment (Lenalidomide, Nivolumab)
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Lenalidomide, Nivolumab) (N=1)
Anemia (Blood and lymphatic system disorders) | 1 (6)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Aspartate Aminotransferasae Increased (Investigations) | 1 (2)
Blood Bilirubin Increased (Investigations) | 1 (2)
Cognitive Disturbance (Nervous system disorders) | 1 (1)
Cough (non-productive) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diarrhea-intermittent (Gastrointestinal disorders) | 1 (1)
Dry Skin- Bilateral Lower Extremities (Skin and subcutaneous tissue disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Eye Hemorrhage (Eye disorders) | 1 (1)
Fatigue (General disorders) | 1 (4)
Generlized Weakness (Musculoskeletal and connective tissue disorders) | 1 (3)
Hip Pain- Bilateral (General disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2)
Insomnia (Psychiatric disorders) | 1 (1)
Localized Edema (Bilateral Ankles) (General disorders) | 1 (1)
Lymphocyte Count Decreased (Investigations) | 1 (1)
Myalgia- Left Rib (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Neutrophil Count Decreased (Investigations) | 1 (1)
Platelet Count Decreased (Investigations) | 1 (5)
White Blood Cell Decreased (Investigations) | 1 (5)

LIMITATIONS AND CAVEATS:
Study was discontinued due to FDA recommendations of the potential toxities of the combination of nivolumab with an immunemodulator(lenalidomide, pomalidomde)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-19): https://cdn.clinicaltrials.gov/large-docs/46/NCT03333746/Prot_SAP_000.pdf